CLINICAL TRIAL: NCT04239235
Title: Comparative Effectiveness of Significant Other-Enhanced OBOT in Primary Care
Brief Title: Integrating Support Persons Into Recovery
Acronym: INSPIRE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Karen Osilla, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-62016
Record Dates: First submitted 2020-01-06; First posted 2020-01-27 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Opioid Addiction
Keywords: Opioid Medication Assisted Treatment; Community Reinforcement Approach and Family Training
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Two-arm RCT where participants are randomly assigned to intervention or control.
Masking Description: Participants will be told which condition they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Community Reinforcement Approach and Family Training is a 10-session rolling group for the support person.
  Interventions: Behavioral: CRAFT
- Control (No Intervention): This condition is for support persons who do not receive CRAFT. They will receive no intervention or usual care services available at the clinic.

INTERVENTIONS:
Behavioral: CRAFT — CRAFT is an evidence-based and non-confrontational approach for teaching friends/family members strategies to help their loved one reduce/refrain from using substances. It focuses on improving the lives of both the friends/family members and the individual struggling with substance use.
  Arms: Intervention

SUMMARY:
INtegrated Support Persons Into Recovery (INSPIRE) is a 4-year research project that tests whether integrating a patient's support person into a patient's treatment with Buprenorphine/Naloxone can improve outcomes. The study will examine whether a counseling program called CRAFT for a support person, such as a family member, spouse or friend, can improve patient outcomes.

DETAILED DESCRIPTION:
Opioid use disorders (OUDs) have reached an all-time high and have devastating effects on the individual, family, and community. While medication treatment for OUD saves lives, rates of treatment drop out are very high. In addition, existing OUD treatments neglect the impact of untreated OUD on the family, and ignore the potential role family members and support persons (SPs) could have on encouraging long-term recovery. Incorporating the patient's support system may be an important way to improve treatment retention. The proposed study evaluates a counseling program for concerned family members, spouses, and friends called Community Reinforcement and Family Training (CRAFT), which is successful at engaging and retaining patients in substance use treatment. While promising, no studies have evaluated whether CRAFT can help patients remain on medication treatment for OUD, provided by community health clinics. If effective, this could save lives and help both patient and family member health outcomes. Patient and SP pairs will be recruited from community health clinics throughout northern and southern California. Patients taking OUD medication treatment will be recruited and randomly assign half of the SPs to receive CRAFT; the other half would receive treatment-as-usual. Patients and SPs will be interviewed three and twelve months later to evaluate whether patients with CRAFT SPs stay in OUD treatment longer, and whether patient and SP health outcomes improve.

ELIGIBILITY:
Patient inclusion criteria:

* 18 and older
* on buprenorphine treatment for OUD
* has an eligible support person that participates

Support person inclusion criteria:

* 18 and older
* frequent contact with the patient
* willing and available to try CRAFT

Patient exclusion criteria:

* < 18 years and older
* not currently receiving buprenorphine
* not able to provide consent

Support person exclusion criteria:

* < 18 years and older
* currently has a problem with heroin or opioid pills
* not able to provide consent
* actively using other substances such that their presence in group would be contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient buprenorphine retention | 6 months after baseline
  Percentage of patients who initiated OBOT who have at least 6 months of continuous treatment with buprenorphine with no more than a 7-day lapse between prescriptions
Patient buprenorphine retention | 12 months after baseline
  Percentage of patients who initiated OBOT who have at least 12 months of continuous treatment with buprenorphine with no more than a 7-day lapse between prescriptions

SECONDARY OUTCOMES:
Patient opioid and other substance use | 3 and 12 months after baseline
  Days of past month use
Patient opioid and other substance use | 3 months after baseline
  Days of past month use
Patient and Support Person depression symptoms | 3 months after baseline
  severity of depression (PHQ-9, Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression)
Patient and Support Person depression symptoms | 12 months after baseline
  severity of depression (PHQ-9, Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression)
Patient and Support Person anxiety symptoms | 3 months after baseline
  severity of anxiety (GAD-7, Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, and severe anxiety)
Patient and Support Person anxiety symptoms | 12 months after baseline
  severity of anxiety (GAD-7, Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, and severe anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Osilla, PhD, Principal Investigator — Stanford University
Locations (6):
- United States (6):
  - Open Door Community Health Centers, Arcata, California
  - Lifelong Medical Care, Berkeley, California
  - Contra Costa Health Services, Concord, California
  - Behavioral Health Services, Gardena, California
  - Family Health Centers of San Diego, San Diego, California
  - Venice Family Clinic, Venice, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osilla KC, Becker K, Ecola L, Hurley B, Manuel JK, Ober A, Paddock SM, Watkins KE. Study design to evaluate a group-based therapy for support persons of adults on buprenorphine/naloxone. Addict Sci Clin Pract. 2020 Jul 11;15(1):25. doi: 10.1186/s13722-020-00199-2. PMID 32653029